CLINICAL TRIAL: NCT01684306
Title: Acute Effects of Modafinil on Brain Resting State Networks in Young Healthy Subjects
Brief Title: Pharmacological Cognitive Enhancement
Acronym: MODREST
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Responsible Party: Principal Investigator, Roberto Esposito, MD,Phd, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MODREST_2011
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Fluid Inteligence; Modafinil; Healthy Young Subjects; Resting State Networks
Keywords: RsfMRI, brain plasticity, cognitive enhancer
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Experimental): Study subjects received, in a double blind fashion, a placebo pill identical to the drug.
  Interventions: Drug: Placebo
- Modafinil (Experimental): Modafinil (Provigil), a drug on the market since 1997, is employed for the treatment of narcolepsy and other sleep disorders. In recent years, modafinil has also been used off-label to treat cognitive dysfunction in psychiatric disorders such as schizophrenia and Attention Deficit/Hyperactivity Disorder (ADHD).
  Study subjects received, in a double blind fashion, either a single dose (100 mg) of modafinil.
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — Study subjects received, in a double blind fashion, either a single dose (100 mg) of modafinil or a placebo pill identical to the drug.
  Other Names: Provigil; Code name: Modafinil; serial number:74507491
  Arms: Modafinil
Drug: Placebo — Study subjects received, in a double blind fashion, either a single dose (100 mg) of modafinil or a placebo pill identical to the drug.
  Arms: Placebo

SUMMARY:
There is growing debate on the use of drugs that can promote cognitive enhancement. Amphetamine-like drugs have been employed as cognitive enhancers, but all of them have important side effects and may induce addiction. In our study, we will investigate the use of modafinil which, in recent years, has been proposed as cognitive enhancer. Modafinil appears to have less side effects compared to amphetamine-like drugs and we will analyzed whether the drug can influence cognitive performances and the brain resting state network activity of healthy young subjects.

DETAILED DESCRIPTION:
Subjects will be included in a double-blind, placebo-controlled study in which a single dose (100 mg) of modafinil will be administered. Both groups will be, before and three hours after administration of drug or placebo, tested for neuropsychological performances with the Raven's Advanced Progressive Matrices II set (APM).

Resting state functional magnetic resonance (rs-fMRI) will be also employed, before and after three hours, to study changes in the activity of resting state brain networks. Finally, with Diffusion Tensor Imaging (DTI) we will evaluate the structural connectivity of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* subjects do not meet the criteria for exclusion

Exclusion Criteria:

* current signs of psychiatric, neurological or medical (hypertension, cardiac disorders, epilepsy) conditions as determined by the Millon test and by clinical examination;subjects showing visual or motor impairments. All subjects taking any psychoactive drug or having a history of alcohol abuse.

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Acute effects of modafinil on brain resting state networks in young healthy subjects | within one week

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neuroscience and Imaging, University "G. d'Annunzio", Chieti, Italy, Italy

REFERENCES:
- [Derived] Cera N, Tartaro A, Sensi SL. Modafinil alters intrinsic functional connectivity of the right posterior insula: a pharmacological resting state fMRI study. PLoS One. 2014 Sep 19;9(9):e107145. doi: 10.1371/journal.pone.0107145. eCollection 2014. PMID 25237810
- [Derived] Esposito R, Cilli F, Pieramico V, Ferretti A, Macchia A, Tommasi M, Saggino A, Ciavardelli D, Manna A, Navarra R, Cieri F, Stuppia L, Tartaro A, Sensi SL. Acute effects of modafinil on brain resting state networks in young healthy subjects. PLoS One. 2013 Jul 25;8(7):e69224. doi: 10.1371/journal.pone.0069224. Print 2013. PMID 23935959